CLINICAL TRIAL: NCT07013994
Title: Comparison of Traditional and Ultrasound-Guided Techniques for Vascular Access in Patients With Difficult Venous Access in Emergency Department: Randomized Clinical Trial Protocol
Brief Title: Comparison of Traditional and Ultrasound-Guided Techniques for Vascular Access in Patients With Difficult Venous Access in Emergency Department.
Acronym: PUVASECO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mercedes Segunda Peralta Gámez (Other)
Collaborators: University Rovira i Virgili (Other)
Responsible Party: Sponsor-Investigator, Mercedes Segunda Peralta Gámez, Graduate in nursing, master's degree in research in nursing sciences., Nuestra Señora de Sonsoles Hospital in Ávila
Organization: Nuestra Señora de Sonsoles Hospital in Ávila (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CAAV/2024/60
Record Dates: First submitted 2025-05-14; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Arterial Blood Pressure; Difficult Vein Access
Keywords: Ultrasonography; Peripheral venous catheter; difficult venous access; arterial blood pressure; nurse

STUDY DESIGN:
Intervention Model Description: Participants who meet the inclusion criteria will be randomly selected to form the control group, which will undergo the traditional technique, and the experimental group, which will undergo the study or ultrasound-guided technique.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Echoguided technique (Experimental): Ultrasound will be used for peripheral venous cannulation and arterial puncture by direct visualisation of the needle in the selected structure.
  Interventions: Procedure: peripheral venous cannulation with ultrasound-guided technique; Procedure: Arterial gas puncture using ultrasound-guided technique
- Traditional technique (Active Comparator): Vascular puncture will be performed using the traditional visualisation/palpation technique.
  Interventions: Procedure: Peripheral venous cannulation with traditional technique; Procedure: Arterial puncture by traditional technique

INTERVENTIONS:
Procedure: peripheral venous cannulation with ultrasound-guided technique — Peripheral venous cannulation with short peripheral vascular access device, performed by ultrasound technique.
  Arms: Echoguided technique
Procedure: Arterial gas puncture using ultrasound-guided technique — Arterial puncture using a needle and heparinised syringe to extract a sample for arterial blood gas analysis, using the ultrasound-guided technique.
  Arms: Echoguided technique
Procedure: Peripheral venous cannulation with traditional technique — Cannulation of a short peripheral vascular access device using the traditional visualisation and palpation technique.
  Arms: Traditional technique
Procedure: Arterial puncture by traditional technique — Arterial puncture using a needle and heparinised syringe to extract an arterial blood sample for arterial gamosetry analysis, performed using the traditional arterial pulse palpation technique.
  Arms: Traditional technique

SUMMARY:
The aim of this clinical trial is to compare the use of ultrasound versus the traditional palpation and visualization technique for vascular punctures, both peripheral venous and arterial punctures for arterial blood gas sampling, in patients presenting to hospital emergency departments. The main questions it seeks to answer are:

Does the use of ultrasound facilitate peripheral venous cannulation in patients with difficult venous access in the emergency department? Does the use of ultrasound facilitate arterial puncture in patients presenting to the emergency department who require arterial blood gases?

The researchers will compare the use of ultrasound with the traditional technique in vascular punctures by emergency department nurses. To determine the differences in the number of attempts needed, the number of professionals needed to perform the technique, the time invested, the pain produced with both techniques, etc., the researchers will compare the use of ultrasound with the traditional technique for vascular punctures by emergency department nurses.

DETAILED DESCRIPTION:
Introduction It is estimated that 90% of patients attending Emergency Departments (ED) require venipuncture, with short peripheral intravenous catheters (PIVC) being the most used invasive devices in healthcare settings. However, there are patients for whom even experienced nurses require more than two attempts to successfully perform the procedure; these patients are classified as having difficult venous access (DIVA). This condition is estimated to occur in 10-24% of adult patients and up to 37% of children. Arterial punctures, often performed to collect blood samples or arterial blood gases (ABG), are similarly common in ED, with first-attempt failure rates reported at approximately 10%.

Failed punctures result in deterioration of the patient's vein and arterial capital, as well as causing pain, stress, and delays in medical care. They also create highly demanding situations for nursing professionals and lead to increased use of human and material resources. To mitigate these issues, certain predisposing factors for DIVA patients have been identified, including obesity, oedema, previous cannulations, and hypotension. Additionally, support tools such as the DIVA scale for pediatric patients and the A-DICAVE scale, validated in 2020 by Dr Salleras, have been developed. The latter is specifically designed for adult patients attending ED. However, no validated scales currently exist for identifying patients at risk of difficult ABG sampling.

Once patients with DIVA are identified, or when difficulties in performing ABG are anticipated, healthcare professionals can employ ultrasound-guided techniques to facilitate these procedures. Ultrasound allows for easier identification of vascular access points, as well as real-time confirmation of puncture success and correct SPVC placement.

Although an increasing number of authors advocate for the use of ultrasound in PIVC placement, existing literature primarily focuses on surgical, anesthetic, or pediatric patients. Consequently, ultrasound-guided techniques are not yet widely adopted, and patients continue to experience the consequences of multiple failed attempts. In the context of ED, studies such as those by Dr Salleras and Rodríguez-Herrera highlight the feasibility and benefits of these techniques. Nevertheless, ultrasound-guided vascular access has not yet been systematically implemented through standardized protocols.

This present study aims to provide evidence on the utility of validated scales for identifying DIVA patients, as well as the benefits of ultrasound-guided vascular punctures in ED. It will consider not only procedural success rates but also the satisfaction of healthcare professionals, patients, and their families.

Hypothesis: The ultrasound-guided puncture facilitates vascular access in patients with difficult vascular conditions, identified using validated scales, who attend Emergency Departments.

Objective: The primary objective of this study is to compare ultrasound-guided techniques with traditional methods for vascular access in DIVA patients identified through validated scales in ED. Additionally, the study will analyze the advantages of incorporating ultrasound-guided techniques into routine clinical practice.

Methodology The study will consist of an open-label RCT to be conducted in Spain, within the ED of a secondary-level hospital. The trial is scheduled to begin in January 2025, with results expected by December 2025.

Design:

The RCT will collect data derived from the procedures performed on patients selected through probabilistic random sampling. The study workflow is outlined in the following flowchart.

Participants The study will recruit DIVA patients identified using the A-DICAVE scale for patients aged >14 years and the DIVA scale for those aged <14 years, who attend the ED and require short PIVC or AGB. Inclusion criteria will include signed informed consent and a score of ≥3 on the A-DICAVE scale or ≥4 on the DIVA scale for PIVC.

Sample Size:

The sample size calculation will be based on the minimum sample size formula for mean comparison. Considering data from a similar study conducted in other healthcare settings and assuming a minimal detectable mean difference of 0.52 and a variance of 1.64 ("number of attempts" variable), a minimum sample size of 95 participants was obtained. Accounting for a 20% loss rate, the required sample size increases to 114 participants, with 57 in each group.

For the sample size required for arterial puncture, the calculation will follow data from a study by Género et al, which reported a 34% difference in success rates using ultrasound compared to the traditional technique. To demonstrate a minimum difference of 37% in first-attempt success rates between the two groups, with an alpha error of 0.5%, 90% power, and accounting for a 20% loss rate, the required sample size is 80 participants, with 40 in each group.

Randomization of the Sample:

Random assignment of participants to the Control Group (CG) and the Experimental Group (EG) will be conducted using a simple randomization method. Each participant will have an equal probability of being assigned to either group, minimizing bias and ensuring the equitable distribution of characteristics between the groups. To achieve this, a computer-generated random number sequence will be used. Additionally, random permuted blocks will be created to reduce the predictability of the random sequence, while ensuring an equal number of subjects in each group.

Details of the sample selection, inclusion criteria applied, and methods used for random assignments to CG and EG will be documented. This will ensure participants' right to withdraw their data and guarantee the transparency and replicability of the study.

Statistical Methods:

The data will be analyzed using SPSS software, version 22. Initially, normality tests will be performed to assess the distribution, homogeneity, and comparability of the sample, employing kurtosis, skewness coefficients, and the Shapiro-Wilk test. A descriptive analysis will then be conducted using measures of central tendency and dispersion (SD) for quantitative variables, alongside calculations of the median and interquartile range (IQR). Qualitative variables will be expressed as frequencies (n) and percentages (%).

Subsequently, appropriate statistical tests will be conducted to determine whether the hypothesis can be rejected, analyzing relationships between the different variables. For qualitative variables, the Chi-square test will be used, or Fisher's exact test if values <5 are observed in the sample. For quantitative variables, the Student's t-test will be applied, or the Mann-Whitney U test in cases where the data do not follow a normal distribution.

In all calculations performed in the study, an alpha error of 0.05 and a beta error of 0.2 will be considered, with a 95% confidence level.

Ethical Considerations:

The study has received approval from the Ethics Committee for Research and Medicines (GASAV/2024/60) and consent from the local healthcare management authorities where the study will be conducted. The research will adhere to the ethical principles outlined in the Declaration of Helsinki and the World Medical Association's six ethical principles for medical research involving human subjects.

The study will comply with the General Data Protection Regulation and Spain's Organic Law 3/2018 on Data Protection, ensuring the confidentiality and anonymity of all participants. The provisions of Law 41/2002 on patient autonomy will also be respected, particularly in cases involving children and patients with cognitive impairments.

Participants will be provided with all necessary information about the study via a Participant Information Sheet and a copy of the informed consent form, which will include the contact details of the principal investigator.

Results Data from the CG will be obtained using the traditional technique, which involves palpation and visualization of veins following the application of a tourniquet to the selected limb for PIVC, and pulse palpation for ABG sampling. For the EG, the ultrasound-guided technique will be employed, beginning with vessel mapping using the RaPeVa technique, identification and measurement of the selected vessel, and an examination of surrounding structures to avoid potential injury. If the practitioner deems it necessary, they may switch techniques, recording the change on the data collection form and accounting for both interventions.

The study design does not allow for blinding of the technique assignment, either for participants or the collaborating nursing professionals. However, an external observer will be responsible for collecting data regarding patient and/or family pain and satisfaction. All data collected will be alphanumerically coded to ensure that analysts remain blinded to the treatment group assignments.

Measurement Instruments

To identify DIVA patients during PIVC catheterization, two scales will be used depending on the patient's age:

* For patients aged ≥14 years, the A-DICAVE scale(11) will be applied. This scale consists of three items: vein visualization (scored 0-2), vein palpation (scored 0-2), and a history of puncture difficulty (scored 0-1). The total score is categorized as follows: easy (0-2 points) and difficult (3-5 points).
* For patients aged <14 years, the DIVA4 scale(21) will be used. This scale scored 0-10, includes four items: visible vein after tourniquet application (0-2 points), palpable vein after tourniquet application (0-2 points), age (≥3 years: 0 points; 1-2 years: 1 point; <1 year: 3 points), and history of prematurity with gestational age <38 weeks (0-3 points). It has been demonstrated that scores >4 typically indicate the need for multiple punctures to achieve adequate venous access.

To assess the satisfaction levels of professionals, patients, and their families, a 5-point Likert satisfaction scale will be applied. If patients are unable to express their satisfaction, only the response from their family members will be recorded.

Pain assessment will utilize numerical scales (0-10):

* For adults and children aged >7 years, the Visual Analogue Scale (VAS)(22) will be used.
* For children aged <5 years, the FLACC scale (Face, Legs, Activity, Cry, Consolability) will be applied.
* For adults with cognitive impairments, the PAINAD scale (Pain Assessment in Advanced Dementia) will be employed.

Data Collection System

Collaborators will be provided with a data collection form accessible at the point of care. A separate form will be used for each technique (PVC or ABG), ensuring that the data are transferred to a dedicated database specifically prepared for the study. The database will record all relevant variables:

Dependent variables Description Type of technique: Arterial puncture, peripheral venous cannulation with short PIVC Total score in the A-DICAVE scale: From 0 to 10 score in patients below 14 Score in DIVA scale: From 0 to 8 score in patients over 14- Score of every item in the A-DICAVE scale: Score of every item in the scale Success Successful result (Yes/No) Number of attempts: Number of punctures attempts to achieve cannulation Numbers of nurses attempting Number of nurses to achieve cannulation Time taken in the technique: Time in minutes taken for the procedure Cannulation zone Pace of insertion of the catheter (hand, forearm, flexure, arm) Catheter gauge: Measurement in gauges of the used catheter Pain: EAV scales (oriented patient), FLACC (pediatric patient) or PAINAD (disorientated patient) Permanence of the vascular access: Permanence time of the catheter Secondary effects Type of effects (extravasation, phlebitis, obstruction, others) Patient satisfaction: Level of satisfaction ( 5-point Likert scale) Family satisfaction: Level of satisfaction of the family (5-point Likert scale) Professional satisfaction: Level of satisfaction of the professional who applied the technique (5-point Likert scale) Independent variables Description Age Years Gender: Male, female, nonbinary Reason of the consultation: Reason for the assistance according to nursing record Emergency zone: Assigned emergency zone Triage level: Classification SET (I , II, III, IV, V) Predisposing factors of DIVA: Factors such as addiction, obesity, old age among others Procedure variables: Description Type of technique: Traditional, ultrasound guided or directed Tube placement: Longitudinal, transversal, none Confusion variables: Description Medication given :Medication used through the access Dilution volume: Volume in ml of the medication dilution Time of administratio:n Taken time in minutes of the administration Conscience level: Glasgow scale Agitation: Yes/No

ELIGIBILITY:
Inclusion Criteria:

* Prescription for CIP or GA cannulation.
* Informed consent signed by the patient or patient's representative.
* A score ≥3 on the A-DICAVE scale or ≥4 on the DIVA scale for PIVC.

Exclusion Criteria:

* Scores below 3 on the A-DICAVE scale or below 4 on the DIVA scale for PIVC.
* Inability to obtain informed consent from the patient or patient's representative

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Scores obtained by DIVA patients on the A-DICAVE scale | At the beginning
  Results of the assessment by the adult patients included in the study using the A-DICAVE scale (Adult Venous Catheterisation Difficulty Scale). With values from 0 to 5. Values greater than or equal to 3 indicate that the patient has difficult venous access.
Scores obtained by DIVA patients on the DIVA scale | At the beginning
  Assessment of paediatric patients using the DIVA scale (Dificil Acceso Vascular). Values above 4 indicate that the patient has a difficult venous access.
Number of patients undergoing successful peripheral venous cannulation | During the intervention, expected time 1 year.
  Successful peripheral venous cannulation using both techniques
Time spent on the techniques to be compared | During the intervention, expected time 1 year.
  Time spent on the techniques from start to completion of the procedure
Number of professionals involved in the technique | During the intervention, expected time 1 year.
  Number of nursing professionals required to perform the technique successfully.

SECONDARY OUTCOMES:
Pain produced by the techniques | During the intervention, expected time 1 year.
  Comparison of the pain perceived by the participants after the techniques, assessed using the validated EVA (Visual analogue scale), FLACC (Face, Legs, Activity, Cry, and Consolabity) and PAINAD scales (Pain Assessment in Advance Dementia). All of them are rated from 0 to 10, with 0 being the absence of pain and 10 being the maximum pain.
Satisfaction perceived by professionals after performing the techniques | During the intervention, expected time 1 year.
  Comparison of the satisfaction perceived by the professionals performing the different techniques under study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Emergency Department of the Nuestra Señora de Sonsoles Hospital in Ávila., Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: No
It is considered that the individual information of the participants will not be relevant, as the information will consist of the variables that allow the comparison of the techniques under study, and these data will be shared with the results. Sharing more information could only violate the protection of participants' privacy without providing relevant data.

REFERENCES:
- [Background] Romo-Miguel P, Ballesteros-Pena S. Ultrasound-guided puncture vs conventional technique for arterial blood gas analysis sampling in adults: A systematic review. Enferm Intensiva (Engl Ed). 2024 Oct-Dec;35(4):368-375. doi: 10.1016/j.enfie.2023.10.003. Epub 2024 Mar 6. PMID 38453623
- [Background] Tran QK, Flanagan K, Fairchild M, Yardi I, Pourmand A. Nurses and Efficacy of Ultrasound-Guided Versus Traditional Venous Access: A Systemic Review and Meta-Analysis. J Emerg Nurs. 2022 Mar;48(2):145-158.e1. doi: 10.1016/j.jen.2021.12.003. Epub 2022 Feb 4. PMID 35125291
- [Background] Salleras-Duran L, Fuentes-Pumarola C, Fontova-Almato A, Roqueta-Vall-Llosera M, Camara-Liebana D, Ballester-Ferrando D. Pain and Satisfaction Perceptions of Ultrasound-Guided Versus Conventional Peripheral Intravenous Catheterization: A Randomized Controlled Trial. Pain Manag Nurs. 2024 Feb;25(1):e37-e44. doi: 10.1016/j.pmn.2023.07.010. Epub 2023 Aug 24. PMID 37633742
- [Background] Osakidetza. Guía de procedimiento de punción arterial para gasometría en población adulta. 2020. Available on: https://www.researchgate.net/publication/339483856_ guia_de_procedimiento_de_puncion_arterial_para_gasometria_en_poblacion_adulta.
- [Background] Kaganovskaya M, Wuerz L. Development of an educational program using ultrasonography in vascular access for nurse practitioner students. Br J Nurs. 2021 Jan 28;30(2):S34-S42. doi: 10.12968/bjon.2021.30.2.S34. PMID 33529109
- [Background] Ocsa C, Gimeno V, Cortés M, Naccarato G, Reinoso G, Nuñez P. Desarrollo de un programa de capacitación en la colocación de catéteres venosos periféricos guiada por ecografía: Experiencia en un hospital pediátrico de tercer nivel. Emerg pediatr. 2024;3(1):44-8.
- [Background] Amick AE, Feinsmith SE, Davis EM, Sell J, Macdonald V, Trinquero P, Moore AG, Gappmeier V, Colton K, Cunningham A, Ford W, Feinglass J, Barsuk JH. Simulation-Based Mastery Learning Improves Ultrasound-Guided Peripheral Intravenous Catheter Insertion Skills of Practicing Nurses. Simul Healthc. 2022 Feb 1;17(1):7-14. doi: 10.1097/SIH.0000000000000545. PMID 33428356
- [Background] McKinney A, Steanson K, Lebar K. A Standardized Training Program in Ultrasound-Guided Intravenous Line Placement: Improving Nurses' Confidence and Success. Adv Neonatal Care. 2023 Feb 1;23(1):17-22. doi: 10.1097/ANC.0000000000000969. Epub 2022 Feb 15. PMID 35170498
- [Background] Rodriguez-Herrera A, Solaz-Garcia A, Molla-Olmos E, Ferrer-Puchol D, Esteve-Claramunt F, Trujillo-Barbera S, Garcia-Bermejo P, Casana-Mohedo J. Use of the Ultrasound Technique as Compared to the Standard Technique for the Improvement of Venous Cannulation in Patients with Difficult Access. Healthcare (Basel). 2022 Jan 29;10(2):261. doi: 10.3390/healthcare10020261. PMID 35206876
- [Background] Lam C, Dunstan L, Sweeny A, Watkins S, George S, Snelling PJ. A survey of paediatric difficult peripheral intravenous access in the emergency department and use of point-of-care ultrasound. Australas J Ultrasound Med. 2023 Jul 13;26(3):184-190. doi: 10.1002/ajum.12353. eCollection 2023 Aug. PMID 37701768
- [Background] Pittiruti M, Van Boxtel T, Scoppettuolo G, Carr P, Konstantinou E, Ortiz Miluy G, Lamperti M, Goossens GA, Simcock L, Dupont C, Inwood S, Bertoglio S, Nicholson J, Pinelli F, Pepe G. European recommendations on the proper indication and use of peripheral venous access devices (the ERPIUP consensus): A WoCoVA project. J Vasc Access. 2023 Jan;24(1):165-182. doi: 10.1177/11297298211023274. Epub 2021 Jun 4. PMID 34088239
- [Background] Salleras-Duran L, Fuentes-Pumarola C, Ballester-Ferrando D, Congost-Devesa L, Delclos-Rabassa J, Fontova-Almato A. Development, Diagnostic Sensitivity, and Prognostic Accuracy of the Adult-Difficult Venous Catheterization Scale for Emergency Departments. J Emerg Nurs. 2020 Nov;46(6):827-837.e2. doi: 10.1016/j.jen.2020.06.013. Epub 2020 Sep 21. PMID 32972765
- [Background] Salleras-Duran L, Fuentes-Pumarola C. [Ultrasound-guided peripheral catheterization]. Enferm Clin. 2016 Sep-Oct;26(5):298-306. doi: 10.1016/j.enfcli.2015.04.002. Epub 2015 Jun 4. Spanish. PMID 26051396
- [Background] Genre Grandpierre R, Bobbia X, Muller L, Markarian T, Occean BV, Pommet S, Roger C, Lefrant JY, de la Coussaye JE, Claret PG. Ultrasound guidance in difficult radial artery puncture for blood gas analysis: A prospective, randomized controlled trial. PLoS One. 2019 Mar 20;14(3):e0213683. doi: 10.1371/journal.pone.0213683. eCollection 2019. PMID 30893349
- [Background] Rodríguez Calero MA, Miquel Rodríguez Calero CA. Definiendo la vía venosa periférica de difícil canalización y los factores de riesgo asociados. Revisión sistemática Defining the venous peripheral via of difficult canalization and risk factors associated. Sistemic review. Medicina Balear. 2019;34(1):12-2018.